CLINICAL TRIAL: NCT03260179
Title: An Open-label Phase Ib, Study, to Determine Safety of Oral AL3810 in Patients With Locally Advanced or Metastatic Gastric, Hepatocellular or Nasopharyngeal Carcinoma
Brief Title: Study to Evaluate the Safety, Preliminary Efficacy and Pharmacokinetics of 3810
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Haihe Biopharma Co., Ltd. (Industry)
Collaborators: Shanghai Institute of Materia Medica, Chinese Academy of Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CL1-80881-008
Record Dates: First submitted 2017-07-20; First posted 2017-08-24 (Actual); Last update posted 2017-08-24 (Actual); Status verified 2017-08

CONDITIONS: Advanced Solid Tumor; Advanced/Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Rabeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- gastric carcinoma (Experimental): 20 gastric carcinoma patients were randomly divided into two groups: 4W on or 3w on/1w off, oral AL3810
  Interventions: Drug: AL3810
- hepatocellular carcinoma (Experimental): 20 hepatocellular carcinoma patients were randomly divided into two groups: 4W on or 3w on/1w off, oral AL3810
  Interventions: Drug: AL3810
- Nasopharyngeal carcinoma (Experimental): 20 Nasopharyngeal carcinoma patients were randomly divided into two groups: 4W on or 3w on/1w off, oral AL3810
  Interventions: Drug: AL3810

INTERVENTIONS:
Drug: AL3810 — Fasting，oral ，4w on or 3w on/1w off
  Arms: gastric carcinoma
Drug: AL3810 — Fasting，oral ，4w on or 3w on/1w off
  Arms: hepatocellular carcinoma
Drug: AL3810 — Fasting，oral ，4w on or 3w on/1w off
  Arms: Nasopharyngeal carcinoma

SUMMARY:
This project intends to make a study of personalized medicine evaluation system establishment for liver cancer, gastric cancer and nasopharynx cancer to provide strong support for the development of Precision Medicine and personalized medicine for the patients of high-incidence-rates cancer in China.

ELIGIBILITY:
Main criteria for inclusion:

1. Adult male or female Chinese subject aged 18 to 70 years, inclusive, at the time of signing the informed consent form, with weight at least 40 kg when screening.
2. Life expectancy ≥ 12 weeks as judged by the Investigator.
3. Histologically or cytologically confirmed, locally advanced or metastatic solid tumor and be limited to:

   * Gastric carcinoma (including gastro-oesophageal junction adenocarcinoma).
   * Hepatocellular carcinoma (Child-Pugh Class A).
   * Undifferentiated nasopharyngeal carcinoma.
4. Each subject should provide at least 5 slides for the formalin fixed and paraffin embedded tumor biopsy (undyed) at the baseline, fresh biopsy or most recent primary tumor sample or metastatic sample is required.
5. Patients, who have progressed on (or not been able to tolerate) standard therapy or for whom no standard anticancer therapy exists.
6. Toxicities from any prior therapy, surgery, or radiotherapy must have resolved to Grade ≤ 1 as per the National Cancer Institute- Common Terminology Criteria for Adverse Events (NCI-CTCAE), excluding alopecia and peripheral neuropathy. For subjects having a prior platinum-based therapy, peripheral neuropathy are required to recover to ≤ CTCAE grade 2.
7. Per RECIST v1.1 guidelines for solid tumors:

   * Patients with gastric carcinoma should have at least one measurable lesion beyond stomach,
   * Patients with Hepatocellular carcinoma and undifferentiated nasopharyngeal carcinoma should have at least one measurable lesion.
8. Adequate bone marrow and organ function as defined by the following laboratory values: (prophylactic use of myeloid growth factors (eg, G-CSF, GM-CSF) is prohibited within 2 weeks before screening)

   * Absolute neutrophil count (ANC) ≥ 1.5x 109/L.
   * Platelet counts ≥ 100 x 109/L.
   * Haemoglobin ≥ 90 g/L (without blood transfusion within the last 2 weeks from screening).
   * Creatinine clearance > 50 mL/min (calculated according to Cockroft-Gault formula).
   * Proteinuria < 1+. If proteinuria ≥ 1+, urine protein quantitation over 24 hours should be < 1.0 g/24hrs.
   * INR ≤ 1.5 and APTT≤ 1.5 Upper Limit of Normal (ULN).
   * AST, ALT ≤ 3 x ULN (≤ 5 x ULN if liver metastases or hepatocellular carcinomas are present).
   * Total Bilirubin < 1.5 x ULN.
   * For Hepatocellular carcinomas patients, albumin ≥ 28 g/dL.
9. Patient has an Eastern Cooperative Oncology Group performance status (ECOG PS) ≤ 1.
10. Patient is able to swallow and retain oral medication.
11. Female subjects, with childbearing potential, has a negative serum pregnancy test at screening (within 7 days of the first investigational product administration). The definition of women with child-bearing potential are defined as "All female subjects after puberty unless they are post-menopausal or not sexually active". Females are considered postmenopausal if they have age-related amenorrhea ≥ 12 consecutive months or if they have undergone hysterectomy or bilateral oophorectomy.
12. Patients who have fully understood the study, and have signed the general Informed Consent Form (ICF) prior to any screening procedures being performed

Main criteria for non-inclusion

1. Patient who has participated in another interventional trial within 28 days prior to starting study medicine. If a subject is joining a non-interventional trial, such as an epidemiological study, or in a survival follow-up period of an interventional trial, he or she may participate in this trial.
2. Expected poor compliance during the study.
3. Patient has symptomatic CNS metastases requiring clinical intervention. The stable patient may participate in this trial, who must have completed any prior local treatment for CNS metastases ≥ 14 days prior to the start of study treatment (including radiotherapy and/or low dose steroid therapy).
4. Patient has a concurrent malignancy or malignancy within 2 years of study enrolment, with the exception of adequately treated and cured non-melanomatous skin cancer, carcinoma in situ of breast and cervix, and superficial bladder cancer.
5. Patient who has received chemotherapy, targeted therapy or immunotherapy within 28 days or ≤ 5 half-lives prior to starting study medicine. Take the longer one. For HCC patient who has received any prior local therapy (hepatic arterial embolization, transcatheter arterial chemoembolization, chemoembolization, radiofrequency ablation, percutaneous ethanol injection or cryoablation) within 4 weeks of starting study medicine •.
6. Previous treatment with Bevacizumab within 3 months of starting AL3810. In addition:

   - Patients with nasopharyngeal carcinoma who received antiangiogenic agent are not allowed.
7. Patients with nasopharyngeal carcinoma located within 5mm of large blood vessels.
8. Patient who has received wide field radiotherapy within 28 days prior to starting study medicine
9. Patient who has received a major surgery within 28 days prior to starting study medicine. The definition of a major surgery refers to grade 3 and 4 surgery specified in <Management of Clinical Practice of Medical Technologies> effective on May 1, 2009 in China,
10. Patient has active cardiac disease or a history of cardiac dysfunction in screening including any of the following:

    * History of documented Congestive heart failure ≥ class II (NYHA New York Heart Association functional classification) or requiring therapy,
    * Ventricular and/or supraventricular arrhythmia requiring therapy;
    * Severe conduction disturbance (including QTc interval prolongation > 450msec [corrected by Fredericia formula], history of severe arrhythmia, or history of familial arrhythmia [e.g., Wolff-Parkinson-White syndrome]),
    * Angina pectoris requiring therapy,
    * Left ventricular ejection fraction (LVEF) < 50% evaluated by cardiac ultrasound (ECHO) or Multi Gated Acquisition Scan (MUGA) ,
    * Uncontrolled arterial hypertension (defined as systolic blood pressure ≥ 140mmHg and/or diastolic blood pressure ≥ 90mmHg with optimized antihypertensive therapy or patients treated with ≥ 2 antihypertensive agents),
    * Hypertension with systolic blood pressure ≥ 160mmHg and/or diastolic blood pressure ≥ 100mmHg with or without antihypertensive therapy.
    * Conduction abnormality requiring a pacemaker or implanted a pacemaker.
11. History of clinically significant or uncontrolled cardiac disease within 6 months prior to starting AL3810, including angina, myocardial infarction, and stroke.
12. Patients with thromboembolic events within 12 months prior to starting AL3810, or at a high risk of such events.
13. Patient with hereditary risks of thromboembolic events.
14. Patient is currently receiving treatment with warfarin or any other oral Anticoagulants
15. Patients with active HBV or HCV infection or known positivity for human immunodeficiency virus (HIV) infection are not allowed. HBV, HCV and HIV will be tested in the screening. Serum HBsAg positive with HBV DNA <104 Copy/mL may participate study. Prophylactic anti-HBV medications application can be accepted. Serum HCV or HIV antibody positive is not allowed.
16. Patients receiving medications known to prolong QTc interval and that may be associated with Torsades de Pointes.
17. Serum potassium (K+) levels below LLN at screening period.
18. Patients who received administration of strong inhibitors of CYP2C8 and/or CYP3A4 or strong inducers of CYP3A4 within 7 days or ≤ 5 half-lives (Take the longer one) prior to starting AL3810. And patient cannot stop taking the medication. .
19. Significant gastrointestinal abnormalities, including ulcerative colitis, chronic diarrhoea associated with intestinal malabsorption, the Crohn's disease, or significant abnormalities decided by investigator. In addition, patients with any grade of gastro-intestinal bleeding events within 3 months prior to starting AL3810 are not allowed.
20. History of grade 3 haemorrhage/bleeding events within 6 months prior to starting AL3810, or history of grade 4 haemorrhage/bleeding events.
21. Known pre-existing clinically significant disorder of the hypothalamic-pituitary axis, thyroid and adrenal gland.
22. Serious/active bacterial, viral or fungal infection requiring systemic treatment.
23. Concomitant uncontrolled severe systemic disease (e.g., uncontrolled diabetes mellitus, uncontrolled ascites, etc.).
24. Psychiatric disorder or altered mental status that would preclude understanding of the informed consent process and/or completion of the necessary study procedures.
25. Known organ dysfunction which would either compromise the patient's safety or interfere with the evaluation of AL3810.
26. Male patients and female patients of child bearing potential unable or unwilling to employ effective contraception (abstinence, barrier method with spermicide, intrauterine device, or steroidal contraceptive for women and barrier method) during the study and for 6 months thereafter.
27. Breastfeeding women.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-08-31 (Estimated); Primary Completion 2019-01-31 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
AE | through study completion, an average of 1 year
  the number of patients with grade 3 and 4 AE according to CTC AE 4.03

SECONDARY OUTCOMES:
ORR | through study completion, an average of 1 year
  The proportion of patients who have observed overall remission (CR) or partial remission (PR) as the overall optimal remission based on the RECIST 1.1.
AUC | up to 3 cycles(28 days/cycle)
  Area under the plasma concentration versus time curve
Cmax | up to 3 cycles(28 days/cycle)
  Peak Plasma Concentration
DoR | through study completion, an average of 1 year
  All patients with the best overall response to CR or PR were required to calculate the duration of the response. This time is the duration (progression or death, whichever occurs first) from the first decision to CR or PR to tumor progression or death (death for any cause)
DCR | through study completion, an average of 1 year
  DCR refers to the percentage of patients who have achieved confirmation during the treatment of CR, confirmed PR and / or SD
PFS | through study completion, an average of 1 year
  To the date of randomization to the date of the onset of the disease or the date of death (regardless of the cause of the death) (whichever is the earlier).

OTHER OUTCOMES:
CD4+/CD8+ | from baseline up to six months(every 8 weeks±7 days )
  cell count of CD4+/CD8+
Growth factor | from baseline up to six months(every 8 weeks±7 days ), C1D15
  the content of growth factor such as VEGF，FGF and PDGF in plasma
Exosomes | from baseline up to six months(every 8 weeks±7 days )
  the content of growth factor such as INFγ and cMyc in plasma

CONTACTS AND LOCATIONS:
Locations (7):
- China (7):
  - The 307th Hospital of Chinese People's Liberation Army, Beijing, Beijing Municipality
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Sun Yat-sen University, Guangzhou, Guangdong
  - The 81st Hospital of People's Liberation Army, Nanjing, Jiangsu
  - Jiangsu Cancer Hospital, Nanjing, Jiangsu
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Sun Yat-sen University Cancer Center, Hangzhou, Zhejiang

REFERENCES:
- [Derived] Zhang Y, Luo F, Ma YX, Liu QW, Yang YP, Fang WF, Huang Y, Zhou T, Li J, Pan HM, Yang L, Qin SK, Zhao HY, Zhang L. A Phase Ib Study of Lucitanib (AL3810) in a Cohort of Patients with Recurrent and Metastatic Nasopharyngeal Carcinoma. Oncologist. 2022 Jun 8;27(6):e453-e462. doi: 10.1093/oncolo/oyab076. PMID 35445718